CLINICAL TRIAL: NCT07272798
Title: Cardiac Self-Efficacy in Patients With Chronic Thromboembolic Pulmonary Hypertension
Acronym: CTEPH3
Status: Recruiting | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Mohammad Bashar Izzat, Professor, Damascus University
Other Study IDs: CTEPH3
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: Chronic thromboembolic pulmonary hypertension; self efficacy; functional capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CTEPH: Patients who are diagnosed with chronic thromboembolic pulmonary hypertension who are eligible for surgical pulmonary thromboendarterectomy

SUMMARY:
This study aims to analyze the effect of Pulmonary Endarterectomy (PEA) on patients' self-confidence in managing their chronic illness.

Patients' confidence (or self-efficacy) will be measured using the following questionnaires: 10-item Perceived Efficacy in Patient-Physician Interaction Scale (PEPPI), Self-Efficacy for Managing Chronic Diseases 6-item Scale (SEMCD-6), Sullivan's cardiac self-efficacy scale 13-items (SCSES). The association between improved confidence and better physical results will be analyzed, such as being able to walk longer (6 mint walk test (6-Minute Walk Test)).

Ultimately, this study will help understanding the psychological side of recovery and might lead to better support programs to help patients feel more capable and live better lives after their operation.

DETAILED DESCRIPTION:
This study specifically focuses on three key domains of self-efficacy relevant to the cardiac patient:

1. Patient-Physician Interaction (PEPPI): Confidence in communication with healthcare providers, which is vital for navigating the complexity of post-operative care, medication management, and identifying emergent issues.
2. Chronic Disease Management (SEMCD-6): Confidence in performing essential self-care tasks, such as managing symptoms, coping with emotional distress, and maintaining a healthy lifestyle.
3. Sullivan's cardiac self-efficacy scale 13-items (SCSES): it focuses on two dimensions: controlling symptoms and maintaining daily function We hypothesize that the successful physical removal of the disease burden via PEA will act as a major "mastery experience," fundamentally boosting a patient's self-efficacy. This improvement is expected to be immediately following the clinical stabilization and persist during follow-up, facilitating better long-term outcomes.

Study Rationale and Novelty

Current literature on CTEPH and PEA is heavily focused on the physiological and hemodynamic aspects of the disease. There is a significant gap in the understanding of the patient-reported psychological factors that contribute to excellent outcomes. This prospective cohort study is unique because:

* It is the first, to our knowledge, to specifically and longitudinally quantify the change in cardiac self-efficacy in patients undergoing PEA.
* It directly links this psychological change to the objective measure of surgical success (change in 6MWT), addressing the secondary objective of determining the correlation between psychological and physiological improvement.
* By using Multiple Linear Regression, the study will identify specific pre-operative baseline factors (e.g., 6MWT) that may predict which patients are most likely to experience a significant post-operative self-efficacy gain or remain at risk for low self-efficacy. This has direct implications for identifying patients who would benefit most from targeted pre-operative psychological support or post-operative rehabilitation strategies.

Expected Impact The findings of this study will contribute significantly to the holistic management of CTEPH patients. If a robust correlation is found between the magnitude of self-efficacy change and improved clinical outcomes or reduced readmission rates, it will provide strong evidence to support the integration of self-efficacy-focused interventions into post-PEA cardiac rehabilitation programs. Ultimately, understanding and bolstering the patient's belief in their ability to manage their condition post-surgery will not only optimize the clinical gains achieved by the PEA but also enhance long-term quality of life and reduce the burden on the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing pulmonary thromboendarterectomy for CTEPH
* Able to read and understand the informed consent form and study questionnaires

Exclusion Criteria:

* Patients undergoing Balloon Pulmonary Angioplasty (BPA) or receiving only medical therapy (as the focus is on the surgical cohort).
* Emergency or salvage PEA procedures (to ensure stable baseline assessment).
* Inability to complete the questionnaires due to severe cognitive impairment, psychiatric illness, or language barrier.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with operable chronic pulmonary thromboembolic pulmonary hypertension undergoing pulmonary thromboendarterectomy
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
10-item Perceived Efficacy in Patient-Physician Interaction Scale (PEPPI) | Preoperatively and 6 months postoperatively
  The scale measures patients perceived self-efficacy. It assesses how confident patients feel in their communication skills with doctors, including explaining health concerns and asking for more information. The scale consists of 10 items where patients rate their confidence on a scale typically from 1 (not at all confident) to 5 (very confident). The total score ranges from 10 to 50, with higher scores indicating higher perceived efficacy.
Self-Efficacy for Managing Chronic Diseases 6-item Scale (SEMCD-6) | Preoperatively and 6 months postoperatively
  This scale measures an individual's confidence in their ability to manage tasks and challenges associated with chronic diseases. It assesses self-efficacy related to managing symptoms, treatment, and the impact of chronic diseases on daily life. The scale includes 6 items where individuals rate their confidence on a numerical scale, typically from 1 ("not at all confident") to 10 ("totally confident"). The responses are averaged to produce a final score. The mean score of the 6 items, ranging from 1 to 10, with higher scores indicating higher self-efficacy.
Sullivan's cardiac self-efficacy scale 13-items (SCSES) | Preoperatively and 6 months postoperatively
  The SCSES measures a patient's confidence in their ability to manage cardiac-related symptoms and maintain daily functioning despite heart disease. The scale assesses cardiac-specific self-efficacy, including two dimensions - control of symptoms (8 items) and maintaining function (5 items). The scale consists of 13 items. Each item asks, "How confident are you that you know or can..." and is rated by patients from 0 ("not at all confident") to 4 ("completely confident"). The scores are summed for a total score. The total score is the sum of 13 items, ranging from 0 to 52, with higher scores indicating higher cardiac self-efficacy.
The 6-minute walk test (6MWT) | Preoperatively and 6 months postoperatively
  The 6MWT measures the functional exercise capacity by assessing the distance a person can walk in six minutes. It evaluates submaximal aerobic capacity, endurance, and overall physical function, particularly useful in cardiopulmonary and chronic disease patients. The patient walks along a flat, straight corridor, ideally 30 meters in length, for 6 minutes. The total distance walked is measured in meters. The test uses a marked corridor with distance markers, a stopwatch, and optionally a pulse oximeter and blood pressure monitor to record physiological responses during the test. Unit of Measurement: Distance walked in meters over 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad B Izzat, FRCS(CTh), Study Director — Damascus University School of Medicine
Locations (1):
- Damascus University Cardiac Surgery Hospital, Damascus, Rif-dimashq Governorate, Syria

IPD SHARING:
Plan to Share IPD: Yes
Data will be deposited in the figshare repository
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be deposited upon completion of study and will be made available permanently
Access Criteria: Open to all

REFERENCES:
- [Background] Blechman EA, Maurice A, Buecker B, Helberg C. Can mentoring or skill training reduce recidivism? Observational study with propensity analysis. Prev Sci. 2000 Sep;1(3):139-55. doi: 10.1023/a:1010073222476. PMID 11525345
- [Background] Andrew CM. Optimizing the human experience: nursing the families of people who die in intensive care. Intensive Crit Care Nurs. 1998 Apr;14(2):59-65. doi: 10.1016/s0964-3397(98)80184-5. PMID 9814208
- [Background] Dardi F, Rotunno M, Guarino D, Suarez SM, Niro F, Loforte A, Taglieri N, Ballerini A, Magnani I, Bertozzi R, Donato F, Martini G, Manes A, Saia F, Pacini D, Galie N, Palazzini M. Comparison of different treatment strategies in patients with chronic thromboembolic pulmonary hypertension: a single centre real-world experience. Int J Cardiol. 2023 Nov 15;391:131333. doi: 10.1016/j.ijcard.2023.131333. Epub 2023 Sep 4. PMID 37673403
- [Background] Fors A, Ulin K, Cliffordson C, Ekman I, Brink E. The Cardiac Self-Efficacy Scale, a useful tool with potential to evaluate person-centred care. Eur J Cardiovasc Nurs. 2015 Dec;14(6):536-43. doi: 10.1177/1474515114548622. Epub 2014 Aug 22. PMID 25149667
- [Background] Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. J Am Geriatr Soc. 1998 Jul;46(7):889-94. doi: 10.1111/j.1532-5415.1998.tb02725.x. PMID 9670878
- [Background] Raguragavan A, Jayabalan D, Dhakal S, Saxena A. A systematic review of the impact of pulmonary thromboendarterectomy on health-related quality of life. Pulm Circ. 2024 Jul 1;14(3):e12407. doi: 10.1002/pul2.12407. eCollection 2024 Jul. PMID 38962182